CLINICAL TRIAL: NCT01912976
Title: A Randomized, Intra-individual, Prospective Study Comparing Methyl Aminolaevulinate Photodynamic Therapy With and Without Er:YAG Ablative Fractional Laser Treatment in Asian Patients With Lower Extremity Bowen's Disease
Brief Title: Study of Methyl Aminolaevulinate Photodynamic Therapy With and Without Er:YAG Laser in Bowen's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A University (Other)
Responsible Party: Principal Investigator, Song Ki-Hoon, Assistant professor, Dong-A University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: DAUDerma-01
Record Dates: First submitted 2013-07-09; First posted 2013-07-31 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Bowen's Disease
Keywords: Bowen's disease; Er:YAG; AFL-assisted; MAL-PDT
MeSH Terms: conditions — Bowen's Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Er:YAG AFL-PDT (Experimental): Right leg on each patients was assigned a single session of Er:YAG AFL-PDT.
  Interventions: Drug: Er:YAG AFL-PDT
- MAL-PDT (Active Comparator): Left leg on each patient was selected to receive 2 sessions of MAL-PDT
  Interventions: Drug: MAL-PDT

INTERVENTIONS:
Drug: Er:YAG AFL-PDT — Er:YAG AFL was performed with 550-600 µm ablation depth, level 1 coagulation, 22% treatment density, and a single pulse. MAL cream was then applied under occlusion for 3 hrs and illuminated with a red light-emitting diode light at 37 J/cm2.
  Other Names: Er:YAG ablative fractional laser-assisted MAL-PDT
  Arms: Er:YAG AFL-PDT
Drug: MAL-PDT — a 1-mm thick layer of MAL (16% Metvix® cream, PhotoCure ASA, Oslo, Norway) was applied to the lesion and to 5 mm of surrounding healthy tissue. The area was covered with an occlusive dressing (Tegaderm, 3M, Saint Paul, MN, US) for 3 hours, after which the remaining cream was removed with saline gauze, and the red fluorescence of porphyrins was visualized with Wood's light. Each treatment area was then separately illuminated with red light-emitting diode (LED) lamps (Aktilite CL128; Galderma, Bruchsal, Germany) with peak emission at 632 nm and total light dose of 37 J cm-2. Areas scheduled to receive MAL-PDT received the second treatment 7 days later.
  Other Names: methyl aminolaevulinate-Photodynamic therapy
  Arms: MAL-PDT

SUMMARY:
Methyl aminolaevulinate photodynamic therapy (MAL-PDT) is an effective treatment for Bowen's disease (BD) of the lower extremities. Er:YAG ablative fractional laser (AFL) treatment removes the stratum corneum to increase MAL uptake and may improve efficacy. However, no studies have directly compared the efficacy of MAL-PDT with and without Er:YAG AFL in treating BD of the lower extremities in Asians.

DETAILED DESCRIPTION:
Bowen's disease (BD) is a form of intraepidermal (in situ) squamous cell carcinoma (SCC) originally described in 1912.1 It presents as a gradually enlarging, well-demarcated erythematous plaque with an irregular border and surface crusting or scaling.2 BD is the frequent precancerous skin lesion in Caucasians.3 In the UK, BD occurrence is most common among patients in their 70s and in women (70-85%), and the majority (60-85%) of cases involve lesions of the lower leg.4,5 BD is estimated to evolve into invasive SCC in 3-5% of cases; therefore, treatment is recommended.6 Current guidelines suggest that the available therapeutic options (including cryotherapy, curettage, excision, topical 5-fluorouracil, and topical imiquimod) are broadly similar in efficacy, with 12-month recurrence rates of approximately 5-10%.7 However, cryotherapy can be painful, making treatment of multiple lesions difficult, and healing can be slow.8 Additionally, topical treatment with 5-fluorouracil or imiquimod is relatively slow and typically causes local irritation.9,10 Photodynamic therapy (PDT) with methyl aminolaevulinate (MAL) is an attractive treatment option for BD with large or multiple patches, and poor healing sites can be treated with good efficacy, low recurrence rates, and good cosmetic outcomes.7 PDT requires light activation of a photosensitizer in the presence of oxygen, which generates reactive oxygen species leading to selective and highly localized destruction of abnormal cells.11,12 MAL is an efficient photosensitizer, with deep lesion penetration resulting from enhanced lipophilicity. Compared to 5-aminolevulinic acid, MAL also has a greater specificity for neoplastic cells.13-15 Because histologic features of BD include full-thickness keratinocyte atypia with disordered maturation, it is typically treated twice within an interval of 1 week.16,17 So, complementary techniques are needed to enhance the penetration and accumulation of MAL in order to improve PDT efficacy and decrease treatment duration.

Er:YAG ablative fractional laser therapy (AFL) can ablate the stratum corneum in a precisely tuned manner without producing significant thermal injury. This approach creates microscopic vertical holes in the ablated tissue, surrounded by thin layers of coagulated tissue.18,19 Since the Er:YAG AFL resurfaces 5-20% of the skin at one time and does not injure the entire thickness of the epidermis, healing times are minimized.18,19 Recent studies have demonstrated that AFL facilitates delivery and uptake of topical MAL deep into the skin, enhancing porphyrin synthesis and photodynamic activation.20,21 The objectives of this study were to compare the efficacy, recurrence rate, cosmetic outcomes, and safety of MAL-PDT with and without the use of Er:YAG AFL in Asian BD patients with multiple lower extremity lesions.

ELIGIBILITY:
Inclusion Criteria:

* Korean patients aged ≥ 18 years who had biopsy-confirmed BD lesions on the lower extremities

Exclusion Criteria:

* porphyria,
* known allergies to the MAL cream or lidocaine,
* pregnancy,
* lactation,
* any active systemic infectious disease,
* immunosuppressive treatment,
* personal history of malignant melanoma,
* tendency towards melasma or keloid formation,
* prior treatment of the lesions within 4 weeks, and
* any indication of poor compliance

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Difference the efficacy between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL-PDT) and standard MAL-PDT. | Efficacy was evaluated at 3 months and 12 months after treatment
  Lesion response was classified as either complete (complete disappearance of the lesion) or incomplete (incomplete disappearance) on the basis of visual examination and palpation. The response of each lesion was clinically evaluated

SECONDARY OUTCOMES:
Difference of the cosmetic outcomes between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL-PDT) and standard MAL-PDT. | Cosmetic outcome was assessed by each investigator for all lesions that achieved a complete response at 3 or 12 months
  It was graded using a 4-point scale: excellent (only slight occurrence of redness or change in pigmentation), good (moderate redness or change in pigmentation), fair (slight-to-moderate scarring, atrophy, or induration), or poor (extensive scarring, atrophy, or induration)

OTHER OUTCOMES:
Difference of the recurrence rates and safety between Er:YAG AFL-assisted MAL-PDT (Er:YAG AFL-PDT) and standard MAL-PDT. | within 12 months after both treatment
  If the case of complete response of lesions, all patients were reviewed at 12 months to check recurrence.
  Adverse events reported by the patient were noted at each follow-up visit, including severity, duration, and need for additional therapy. All events due to PDT were described as phototoxic reactions (i.e. erythema, postinflammatory hyperpigmentation, oedema, itching, oozing, bleeding, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Ki-Hoon Song, M.D., Ph.D., Study Chair — Assistant professor and Chariman, Department of dermatology Dong-A University, College of medicine
Locations (1):
- Dong-A University, Busan, Dong Dae Sin-dong, Seo-gu, South Korea